CLINICAL TRIAL: NCT04831931
Title: The Effectiveness of the Exercise Program Applied by Telerehabilitation Method in Individuals With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, merve özel, physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C92F2628X5
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Neck Pain
Keywords: Neck pain, telerehabilitation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised Exercise Group (Experimental): Telerehabilitation will be applied in this group, which will last 4 weeks, and include the following processes
  * Exercises that will be performed every Monday will be taught and applied face-to-face under the supervision of the therapist with online videoconferencing method. Then, videos of weekly exercises that will be prepared by the therapist will be transmitted online to patients.
  * Patients will be asked to perform these exercises 4 days a week in the same week, on Wednesdays, Fridays and Sundays.
  * Also, a video call will be made on Fridays to evaluate whether the movements are done effectively and correctly, and questions of patients (if any) will be answered.
  * Patients will be informed by the physiotherapist that they should send messages on Wednesdays and Sundays to show that they are doing the exercises.
  * The exercise program of new week will be taught every Monday for 4 weeks, the prepared video will be sent, and the program will be advanced and completed.
  Interventions: Other: Exercise Program Applied by Telerehabilitation
- Exercise Group (Active Comparator): Exercise recommendations will be made to this group. Videos and photographs of weekly exercises prepared by the therapist will be sent online to the patient every Monday for 4 weeks, patients will be advised to repeat these exercises 4 days a week.
  Interventions: Other: Exercise Program Applied by Telerehabilitation
- Control Group (No Intervention): No exercise application will be done in this group.Evaluation tests will be applied for 4 weeks only online.

INTERVENTIONS:
Other: Exercise Program Applied by Telerehabilitation — Patients will be evaluated 3 times for 4 weeks throughout the study; before the study commences, at the end of 2th and 4th week
  Exercises will be planned to last for 15 minutes a day, and will be progressed and changed weekly throughout the study period. To the exercise program; It will be created as a progressive program by including stretching, normal range of motion movements, neck, core and scapular stabilization and strengthening exercises and the same program will be given to both groups.
  Arms: Exercise Group; Supervised Exercise Group

SUMMARY:
Neck pain is a common musculoskeletal problem occurring as one of the first conditions causing decreased quality of life and disability.

An estimated 67.5% of people experience neck pain in their lives (5, 6). When the adult population is considered (15-74 years old), the prevalence ranges from 5.9% to 38.7%.

Causes of neck pain are largely variable, and include working in unsuitable ergonomic positions, sitting for a long time, and keeping the neck in abnormal physiological position for a long time.

Various factors are effective in the chronic stage of neck pain. Neck pain is associated with decreased strength and endurance of the cervical muscles. It was observed that deep flexor muscles are weak and superficial flexor muscle activity is increased in patients with neck pain; and that exercise is effective in reducing neck pain because strength, endurance, and flexibility can be regained in the structures around the damaged tissue.

There are several approaches that were found to be effective in the treatment of neck pain. These treatment strategies include physical therapy modalities, manual therapy, therapeutic exercise (stretching, strengthening, and endurance exercises) and home exercise programs.

Home exercise programs are used to expand the clinic-based physical therapy approaches to treat neck pain.

It was stated that it is now compulsory to develop new rehabilitation models and practices to cope with global increase in elderly population, limited resources allocated to public health, and changes in population needs. Telerehabilitation is recommended as a solution to provide physical therapy services; however, it was reported in previous studies that more studies are required in this field to accept its effectiveness.

The purpose of the present study is to examine the effects of 4-week exercise protocol established with stretching, strengthening the scapula muscles for the neck and upper body, neck and core stabilization exercises by ensuring the follow-up of the patients with Telerehabilitation Method on patients' neck pain, Daily Life Activities (DLA), and quality of life by comparing its effects with individuals who apply only home program.

ELIGIBILITY:
Inclusion Criteria:

* voluntary individuals suffering from neck pain for at least 3 months
* over the age of 18
* have a minimum score of 3/10 according to the Numeric Pain Rating Scale
* who fill out the pain preliminary information form, and who will agree to participate in the study through this form.

Exclusion Criteria:

* Pregnant women,
* History of malignancy
* Congenital deformities or surgery history in the neck or shoulder area
* perception problems for verbal commands
* not having internet access
* not having equipment to make video calls

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  Numeric Pain Rating Scale (NPRS) will be used to evaluate pain subjectively. NPRS is used to evaluate pain. The patient is asked to rate the severity of pain over 10, 0 showing no pain, and 10 showing the worst pain score. Validity and validation of the use of NPRS to evaluate chronic pain in the literature with face-to-face and telepresentation methods.
  Its reliability has been reported
Deep Neck Flexor Endurance Test | 4 weeks
  Patients are asked to lie on a flat ground in the form of a "hook" during the online video conference. They are then asked to move their jaws closer to their chests in the Chin Tuck Position, raise their heads approximately 2.5 cm, and remain in this position. If patients experience any pain and fatigue or put their heads back on the floor, the test is terminated. The physiotherapist keeps track of the patient during this period. Two measurements are made, and the long-lasting result is recorded. The validity and reliability of the evaluation has been demonstrated by the online video videoconferencing method.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | 4 weeks
  The level of disability associated with the neck pain will be evaluated with the Neck Disability Index. The NDI consists of 10 sections that include pain sensitivity, personal care, weight lifting, reading, headaches, concentration, work/job, driving, sleep, and social activities. Each question has 6 answer options measuring the severity of pain or limitation. Scoring is done between 0 and 5. The highest score is 50, and the minimum score in 0.
  According to the total score; 0-4 means no limitation, 5-14 means slight limitation, 15-24 moderate limitation, 25-34 severe limitation, 34 and above completely limitation . The Turkish validity and reliability study of the survey was conducted.
World Health Organization Quality of Life Scale-Short Form (WHOQOL-Bref) | 4 weeks
  There are two versions of this scale as the long (WHOQOLS-100) and short (WHOQOLS-27) form. The scale measures the bodily, spiritual, social, and environmental well-being of the individual, and consists of 26 questions. The Turkish version consists of 27 questions. The 27th question is the national question determining the Environmental Area Score. The scale can be applied to non-elderly adults . The field scores are calculated between 4 and 20 because each field refers to the quality of life in the relevant field independently from each other. As the score increases, the quality of life increases. The Turkish validity and reliability study of the scale was conducted .

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makela M, Heliovaara M, Sievers K, Impivaara O, Knekt P, Aromaa A. Prevalence, determinants, and consequences of chronic neck pain in Finland. Am J Epidemiol. 1991 Dec 1;134(11):1356-67. doi: 10.1093/oxfordjournals.aje.a116038. PMID 1755449
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Cohen SP, Hooten WM. Advances in the diagnosis and management of neck pain. BMJ. 2017 Aug 14;358:j3221. doi: 10.1136/bmj.j3221. PMID 28807894
- [Background] May S, Gardiner E, Young S, Klaber-Moffett J. Predictor Variables for a Positive Long-Term Functional Outcome in Patients with Acute and Chronic Neck and Back Pain Treated with a McKenzie Approach: A Secondary Analysis. J Man Manip Ther. 2008;16(3):155-60. doi: 10.1179/jmt.2008.16.3.155. PMID 19119405
- [Background] Peterson C, Bolton J, Humphreys BK. Predictors of outcome in neck pain patients undergoing chiropractic care: comparison of acute and chronic patients. Chiropr Man Therap. 2012 Aug 24;20(1):27. doi: 10.1186/2045-709X-20-27. PMID 22920497
- [Background] Christensen JO, Knardahl S. Time-course of occupational psychological and social factors as predictors of new-onset and persistent neck pain: a three-wave prospective study over 4 years. Pain. 2014 Jul;155(7):1262-1271. doi: 10.1016/j.pain.2014.03.021. Epub 2014 Apr 2. PMID 24704365
- [Background] Ylinen J. Physical exercises and functional rehabilitation for the management of chronic neck pain. Eura Medicophys. 2007 Mar;43(1):119-32. PMID 17369784
- [Background] Moffett J, McLean S. The role of physiotherapy in the management of non-specific back pain and neck pain. Rheumatology (Oxford). 2006 Apr;45(4):371-8. doi: 10.1093/rheumatology/kei242. Epub 2005 Dec 6. PMID 16332949
- [Background] Zronek M, Sanker H, Newcomb J, Donaldson M. The influence of home exercise programs for patients with non-specific or specific neck pain: a systematic review of the literature. J Man Manip Ther. 2016 May;24(2):62-73. doi: 10.1179/2042618613Y.0000000047. PMID 27559275
- [Background] Hailey D, Roine R, Ohinmaa A, Dennett L. Evidence of benefit from telerehabilitation in routine care: a systematic review. J Telemed Telecare. 2011;17(6):281-7. doi: 10.1258/jtt.2011.101208. Epub 2011 Aug 15. PMID 21844172
- [Background] Rogante M, Grigioni M, Cordella D, Giacomozzi C. Ten years of telerehabilitation: A literature overview of technologies and clinical applications. NeuroRehabilitation. 2010;27(4):287-304. doi: 10.3233/NRE-2010-0612. PMID 21160118
- [Background] Galea MD. Telemedicine in Rehabilitation. Phys Med Rehabil Clin N Am. 2019 May;30(2):473-483. doi: 10.1016/j.pmr.2018.12.002. Epub 2019 Mar 5. PMID 30954160
- [Result] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Result] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Result] Mani S, Sharma S, Singh DK. Concurrent validity and reliability of telerehabilitation-based physiotherapy assessment of cervical spine in adults with non-specific neck pain. J Telemed Telecare. 2021 Feb;27(2):88-97. doi: 10.1177/1357633X19861802. Epub 2019 Jul 4. PMID 31272309
- [Result] Edmondston SJ, Wallumrod ME, Macleid F, Kvamme LS, Joebges S, Brabham GC. Reliability of isometric muscle endurance tests in subjects with postural neck pain. J Manipulative Physiol Ther. 2008 Jun;31(5):348-54. doi: 10.1016/j.jmpt.2008.04.010. PMID 18558277
- [Result] Sebastian D, Chovvath R, Malladi R. Cervical extensor endurance test: a reliability study. J Bodyw Mov Ther. 2015 Apr;19(2):213-6. doi: 10.1016/j.jbmt.2014.04.014. Epub 2014 Apr 18. PMID 25892374
- [Result] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Result] Bicer A, Yazici A, Camdeviren H, Erdogan C. Assessment of pain and disability in patients with chronic neck pain: reliability and construct validity of the Turkish version of the neck pain and disability scale. Disabil Rehabil. 2004 Aug 19;26(16):959-62. doi: 10.1080/09638280410001696755. PMID 15371043
- [Result] Aydemir Ö., Köroğlu E., Psikiyatride Kullanılan Klinik Ölçekler. 3'üncü baskı. Ankara. Hekimler Yayın Birliği , 2007; 346-353
- [Result] Eser E, Fidaner H, Fidaner C, Eser SY ve ark. Psychometric properties of WHOQOL-100 and WHOQOL-BREF. 3P Dergisi 1999;7(2 Suppl.):23-40
- [Result] Eser SY, Fidaner H, Fidaner C, Elbi H ve ark. Measure of quality of life WHOQOL-100 and WHOQOL-Bref. 3P Dergisi 1999;7(2 Suppl.):5-13.